CLINICAL TRIAL: NCT03748173
Title: Infasurf®(Calfactant) Aerosol for Infants With Bronchiolitis-AERO-04 A Pilot Study of Aerosol Surfactant for Bronchiolitis in Infants
Brief Title: Infasurf®(Calfactant) Aerosol for Infants With Bronchiolitis-AERO-04
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slowdown due to covid
Sponsor: ONY (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aero-04
Record Dates: First submitted 2018-11-15; First posted 2018-11-20 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — calfactant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): Subjects randomized to the aerosol surfactant evaluation will occur at the end of 60 minutes, with the aerosol continued if the bronchiolitis score is > 4 or there has been less than a 2-point improvement in the bronchiolitis score. Similar evaluation will be performed, if necessary, at 30-minute intervals (maximum 2 hours) with stoppage of the aerosol for an improved bronchiolitis score (≤ 4 or 2-point improvement) at any of the time points. The aerosol would be stopped at any time for significant sustained deterioration in clinical status or any serious adverse event felt related to the treatment. Retreatment can be given at > 4 but < 24 hours if the initial response was positive and there has been subsequent deterioration.
  Interventions: Combination Product: Aerosolized Infasurf
- Usual Care (No Intervention): The only difference in care between treatment and usual care will be treatment with up to two doses of aerosolized Infasurf®.

INTERVENTIONS:
Combination Product: Aerosolized Infasurf — Infants randomized to aerosol treatment will receive Infasurf® aerosol at a rate of 12 ml/hour (the maximal rate using the Solaris CAG). The initial treatment will be for 60 minutes, with reevaluation every 30 minutes thereafter, with a maximum dose of 6 mL/Kg body weight or 2 hours of aerosolization. Treatment will be stopped after 60 minutes (and subsequently at 30-minute intervals) if a 2 point reduction in bronchiolitis score or a score ≤ 4 is achieved. Treatment will also be stopped at any time should there be evidence of other-than-transient deterioration in oxygenation or clinical status or for any serious adverse effect deemed by the infant's clinician to be possibly related to the drug administration.
  Other Names: Calfactant
  Arms: Treatment

SUMMARY:
Delivery of aerosolized Infasurf to bronchiolitis patients with who are not on assisted ventilation can provide sufficient delivery of Infasurf to small airways to improve ventilation and thereby shorten the duration of the respiratory illness.

DETAILED DESCRIPTION:
This pilot clinical trial will compare "usual care" to aerosolized Infasurf. The study objective is to determine

1. Do bronchiolitis patients tolerate aerosolized Infasurf?
2. Does aerosolized Infasurf induce an improvement in respiration?
3. If it does how large a dose is required to observe a positive effect?
4. Is the positive effect transient, if so what is the range of duration of the effect?
5. Does retreatment also result and a positive response?
6. Does aerosolized Infasurf result in more rapid sustained improvement? is superior to.

ELIGIBILITY:
Inclusion Criteria:

1. Infant ≤ 4 months of age admitted to the PICU with the clinical diagnosis of bronchiolitis
2. Severe illness as reflected by a bronchiolitis score ≥ 4 and requiring high flow nasal cannula or continuous positive airway pressure for respiratory support
3. Within 4 hours of PICU admission.

Exclusion Criteria:

1. Need for non-invasive BiPAP or invasive ventilation
2. Significant Co-morbidities

   1. Chronic lung disease (evidenced by supplemental oxygen, home ventilation, or chronic diuretic therapy for CLD)
   2. Unrepaired congenital heart disease
   3. Immune compromise
   4. Neuromuscular weakness
3. Tracheostomy
4. Influenza as the etiologic agent of bronchiolitis
5. Inability to stabilize the infant to a bronchiolitis score < 8

Ages: 0 Months to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Improvement in Respiratory Status | 24 hours post PICU admission
  Incidence of positive respiratory response to Infasurf® Aerosol defined as Bronchiolitis Clinical Score decreased by 2 points or to ≤4.

SECONDARY OUTCOMES:
Need of Respiratory support | 24 hours post PICU admission
  Incidence of need for non-invasive (BiPAP, NIV-NAVA) or invasive ventilation

OTHER OUTCOMES:
Dose as Measured as duration of the therapy | 24 hours post PICU admission
  To determine the optimal dose/duration of aerosolized Infasurf® in infants with bronchiolitis by aerosolizing Infasurf at 35mg/ml at a rate of 1.8 to 2.2 mls per minute until therapeutic response is achieved or the maximum amount of a single dose is reached.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Richmond at VCU, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No